CLINICAL TRIAL: NCT04142554
Title: Window of Opportunity Study of Parsaclisib in Subjects With Newly Diagnosed Stage I-IIIC Triple-Negative or HER2-Positive Breast Cancer
Brief Title: Parsaclisib in Newly Diagnosed Stage I-IIIC Triple Negative or HER2+ Breast Cancer
Acronym: LCCC1820
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn from funding source.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC1820
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Breast Neoplasms; Triple Negative Breast Cancer; HER2-positive Breast Cancer
Keywords: breast; triple negative; HER2-positive; parsaclisib
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm: Parsaclisib ( Dose De-Escalation ) (Experimental): Prior to their scheduled standard of care surgery or research biopsy, subjects (n = 5 per dosing cohort) will be given oral doses of parsaclisib (10, 3.0 or 1.0 mg) once daily over 14 consecutive days.
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib tablets (1.0, 2.5 or 5 mg) are administered orally daily for up to 14 days

SUMMARY:
The purpose of this research study is to find the lowest dose of the cancer drug parsaclisib that has an effect on the type of breast cancer a participant has. Researchers are looking at how Parsaclisib affects the immune system. They want to learn whether and how it helps the immune system to find cancer cells to fight them.

Parsaclisib is an oral drug that limits the effects of a protein called phosphatidylinositol 3-kinase δ (PI3K). By limiting P13K, parsaclisib can block certain cells that prevent the immune cells from working. As a result, it may help the body's immune system to fight tumors. Parsaclisib is being studied in several clinical trials to treat different types of cancers. Parsaclisib has not yet been approved by FDA for the treatment of cancer.

Studies have shown that a good way to find out how cancer acts when exposed to anti-cancer drugs is through a pre-operative window study. In this type of study, tissue and blood are collected before treatment. Then subjects receive a study drug for a few weeks before surgery. Blood is drawn during the course of treatment, and leftover tissue is collected during surgery. Comparing the tissue and blood before and after treatment shows the effects the study drug may have had on the tumor.

Research shows that cancers differ when you look at the DNA and RNA (genetic codes) that are inside a cancer cell. DNA and RNA carry genetic information that can determine traits in humans (such as eye color, height, reaction to treatment, etc.), as well as the traits of cancer cells. Depending on the genetic profile (particularly DNA and RNA) of the cancer, it may respond differently to parsaclisib. In this study, the investigators will look at the genetic profile of a participant's tumor by studying tissue and blood samples collected before and after receiving treatment.

DETAILED DESCRIPTION:
Surgery and Treatment:

Subjects must consent to having tissue collected for research purposes during a pre-treatment research biopsy, and scheduled surgery or end of treatment research biopsy prior to study entry. Prior to their scheduled standard of care surgery or research biopsy, subjects (n = 5 per dosing cohort) will be given oral doses of parsaclisib (10, 3.0 or 1.0 mg) once daily over 14 consecutive days. Cohorts will be enrolled sequentially by dose, where the cohort with the highest dose will be enrolled first and then the next cohort with the next highest dose will be enrolled after the enrollment of the prior cohort completes.

At each dose level it will be determined whether either a 50% increase in the intratumoral CD8+ T cells/regulatory T- cell ratio or a 50% decrease in the intratumoral percentage of regulatory T cells is observed in at least 3 subjects out of 5 at that dose level. If this criterion is met, enrollment in the next highest dose level will commence. This procedure will be repeated until either this criterion is met at the lowest dose level, or when the criterion is not satisfied in a particular dose level. In the latter case, the next highest dose level will be chosen as the "minimum effective dose". In the former case, the lowest dose level will be chosen as the minimum effective dose. The doses being administered are lower than the therapeutic dose levels of parsaclisib (i.e., 20 to 30 mg once daily) recommended for subjects with lymphoma. If the criterion is not met in the first (highest) dose level, then the investigators assume the minimum effective dose is the therapeutic dose of parsaclisib (20 mg once daily) and the study will be terminated.

Blood samples will be collected prior to parsaclisib treatment for research purposes. Subjects will undergo their standard of care surgical procedure or research biopsy within 72 hours (preferably within 24 hours) of completing drug treatment. Tissue and blood samples will be collected for correlative studies during surgery or during a research biopsy procedure. Subjects who have at least 7 days of parsaclisib treatment will be considered evaluable and may have tissue collected even if they have not completed the entire 14 day treatment regimen.

Duration of Follow Up:

Subjects will be followed post-operatively as per routine standard of care. Contraceptive use should continue for 93 days after the last dose of study drug administration. Subjects removed from study treatment for unacceptable adverse events will be followed until resolution or stabilization of the adverse event. Monitoring for AEs should continue for at least 30 days after the last dose of parsaclisib is administered. AEs related to therapy will then be followed until resolution to grade ≤1, or until the condition has stabilized with no further change expected.

ELIGIBILITY:
Inclusion Criteria:

* Is able to understand and give written informed consent for removal of at least 2 cores of tissue via a pre-treatment research biopsy. Is able to understand and give written informed consent for either collection of leftover tissue at time of surgery and via an end of treatment (EOT) research biopsy).
* Is ≥ 18 years of age.
* Has histologically confirmed newly diagnosed Stage I-IIIC invasive breast cancer that is triple negative (ER/PR <1%, HER2 negative) or HER2-positive, and meets the criteria listed below:

  a. HER 2 positive or overexpressed HER2 confirmed by immunohistochemistry (IHC), and florescence in situ hybridization (ISH) according to the 2018 ASCO-CAP guideline: i. IHC score of 3+ without ISH HER2/CEP17 OR ii. ISH HER2/CEP17 amplified with ratio higher than 2.0 OR if reported average HER2 copy number ≥ 6 signals/cell b. Scheduled for lumpectomy, mastectomy or neoadjuvant chemotherapy as first treatment for cancer c. No prior or current therapy for breast cancer d. Amenable to a baseline research breast biopsy e. Amenable to a post-therapy research biopsy (for patients going on to neoadjuvant chemotherapy and not straight to surgery). For patients going directly to surgery, post-therapy biopsy will be obtained at the time of surgery.
* Must have sufficient time to receive at least 7 consecutive days of parsaclisib therapy prior to definitive surgery or initiation of chemotherapy..
* Has an ECOG performance status ≤ 1.
* Is able to swallow and retain oral medication.
* Demonstrates adequate organ function as defined below; all screening labs to be obtained within 72 hr of initiating study treatment.

  1. Hemoglobin (Hgb) - ≥ 10.0 g/dL
  2. Absolute Neutrophil Count (ANC) - ≥ 1.5 × 109/L
  3. Absolute Lymphocyte Count (ALC) - >500 cells/μL
  4. Platelets - ≥ 100 × 109/L
  5. Creatinine - ≤1.5 × ULN OR Calculated creatinine clearance - ≥ 60 mL/min for subject with creatinine levels > 1.5 × ULN (creatinine should be calculated per institutional standard)
  6. Bilirubin - ≤ 1.5 × ULN or direct bilirubin ≤ ULN for subject with total bilirubin >1.5 × ULN
  7. Aspartate aminotransferase (AST) - ≤ 2.5 × ULN
  8. Alanine aminotransferase (ALT) - ≤ 2.5 × ULN
  9. Albumin - ≥2.5 g/dL
  10. International Normalized Ratio (INR) or Prothrombin Time (PT) and Activated Partial Thromboplastin Time (aPTT) - ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT and PTT is within therapeutic range of intended use of anticoagulants
* As determined by the enrolling physician or protocol designee, the subject is able to understand and comply with study procedures.
* For female subjects of childbearing potential: has a negative serum pregnancy test at screening within 72 hours of receiving study treatment. In addition, female subjects must either:

  1. Agree to the use of an approved method of contraception (i.e., two adequate barrier methods throughout the study starting with the screening visit) and to continue its use for the duration of the study treatment through 30 days after the last dose of parsaclisib if a female subject of child-bearing potential, or
  2. Has documented inability to become pregnant (e.g., hysterectomy, bilateral tubal ligation or oophorectomy, or post-menopausal as defined as total cessation of menses for 2 years). Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure otherwise the subject must be willing to use 2 adequate barrier methods throughout the study.

Exclusion Criteria:

* Prior history of another known malignancy other than breast cancer within the previous 2 years with the exception of adequately treated basal cell carcinoma or cervical intraepithelial neoplasia, cervical carcinoma in situ or melanoma in situ.
* Is pregnant or lactating.
* Has a concomitant medical condition that precludes adequate study treatment compliance or assessment, such as bleeding disorders or any other medical condition that would increase risks of additional core biopsy for biomarkers.
* Use of any potent CYP3A4 inhibitors or inducers (e.g., grapefruit or grapefruit juice) within 14 days or 5 half-lives (whichever is longer) before the first dose of parsaclisib.
* Has allergy to inactive components of the study medication.
* History of autoimmune disease or irritable bowel syndrome (IBS), or active colitis.
* Inability to take oral medications (e.g., impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral medications such as ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Is participating in another therapeutic clinical trial or has received another investigational agent within 30 days prior to informed consent.
* Known Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which is allowed).
* Has acute or currently active/requiring anti-viral therapy, hepatic or biliary disease (with the exception of subjects with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Medical history of a disease that requires ongoing steroid therapy for >14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Minimum effective dose of parsaclisib | At time of surgery (2 weeks after start of parsaclisib)
  To determine the minimum dose of parsaclisib, administered once daily for 14 consecutive days, needed in subjects with triple-negative or human epidermal growth factor receptor 2 (HER2) positive breast cancer to result in either a 50% increase in the intratumoral cluster of differentiation 8 (CD8+) Thymus (T) cells/regulatory T cell ratio or a 50% decrease in the percentage of intratumoral regulatory T cells as measured using single cell transcriptomics and/or flow cytometry.

SECONDARY OUTCOMES:
Minimum dose of parsaclisib needed to decrease peripheral blood regulatory T cells | At time of surgery (2 weeks after start of parsaclisib)
  To determine the minimum dose of parsaclisib, administered once daily for 14 consecutive days, in subjects with triple-negative or HER2 positive breast cancer resulting in either a 50% increase in the peripheral blood CD8+ T cells/regulatory T-cell ratio or a 50% decrease in the percentage of peripheral blood regulatory T cells as measured using single cell transcriptomics and/or flow cytometry.
Changes in regulatory T cell signature | At time of surgery (2 weeks after start of parsaclisib)
  To identify changes in the regulatory T cell signature following treatment with parsaclisib in subjects with triple-negative or HER2-positive breast cancer. A regulatory T-cell gene signature expression score is defined as the average of upper quartile normalized and log2 transformed gene expression values of all genes belonging to that gene signature was calculated for each sample. Gene expression values will be determined via RNA-sequencing. A one-sided paired t-test will be used to test for significant pre-post reductions in signature values in each subject, reflecting a decrease in the abundance of intratumoral regulatory T cells.
Changes in Ki-67 mRNA expression | At time of surgery (2 weeks after start of parsaclisib)
  To identify changes in Ki-67 messenger Ribonucleic acid (mRNA) expression following treatment with parsaclisib in subjects with triple-negative or HER2-positive breast cancer. Ki-67 expression pre versus post treatment will be assessed using the average log2 fold change in gene expression between conditions.
Comparison of reduction in the regulatory T cell signature by dose of parsaclisib | At time of surgery (2 weeks after start of parsaclisib)
  The reduction in the regulatory T cell signature by dose of parsaclisib (10 mg, 3.0 mg or 1.0 mg) will be measured as Pre and post-treatment levels of regulatory T-cell total abundance (cell count) and relative abundance (percentage of all cells), and change in relative abundance (fold change in % abundance post vs pre-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Carey Lisa, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials